CLINICAL TRIAL: NCT01088633
Title: Characterization of Aerosol Generation and Transport in the Human Lung of Subjects With Chronic Obstructive Pulmonary Disease
Brief Title: Characterization of Aerosol Generation and Transport in the Human Lung of Subjects With Chronic Obstructive Pulmonary Disease (COPD)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fraunhofer-Institute of Toxicology and Experimental Medicine (Other)
Responsible Party: Principal Investigator, Prof. Dr. Jens Hohlfeld, MD, Division director, Fraunhofer-Institute of Toxicology and Experimental Medicine
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Basic Science
Other Study IDs: 10/05 AEROC
Record Dates: First submitted 2010-03-12; First posted 2010-03-17 (Estimated); Last update posted 2023-09-14 (Actual); Status verified 2023-09

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Exhaled particle analysis (Other)
  Interventions: Other: Exhaled particle analysis

INTERVENTIONS:
Other: Exhaled particle analysis — At visit 2, the exhaled particle analysis will be performed. Subjects will be asked to breath through the device and to perform several breathing maneuvers such as deep breathing, shallow breathing, rapid breathing, slow breathing. These measurements will be repeated after 2 hours on the same day.
  Visit 3:
  After a baseline exhaled particle analysis, the subjects will inhale nebulized saline (2.5 ml of a 0.9 % NaCl-solution). Aerosol generation and transport will be recorded immediately after the end of inhalation as well as 2 hours and 4 hours after the start of inhalation using the same techniques as in visit 2.

SUMMARY:
This study is aiming at evaluating the characteristics of particle emission in subjects with different stages of chronic obstructive pulmonary disease (COPD) compared with healthy smokers.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female subjects, aged ≥ 18 years
2. COPD: Physician diagnosis of chronic obstructive pulmonary disease (COPD GOLD I to IV according to GOLD guidelines)9
3. Healthy smokers: current smokers with a history of at least 10 packyears and no signs of bronchial obstruction in spirometry (FEV1 >= 80% pred, FEV1/FVC >= 70%)
4. Able and willing to give written informed consent
5. Women will be considered for inclusion if they are:

   * not pregnant, as confirmed by pregnancy test, and not nursing
   * of non-child bearing potential (i.e. physiologically incapable of becoming pregnant, including any female who is pre-menarchial or post-menopausal, with documented proof of hysterectomy or tubal ligation, or meet clinical criteria for menopause and has been amenorrhoeic for more than 1 year prior to the screening visit)
   * of childbearing potential and using a highly effective method of contraception during the entire study (vasectomized partner, sexual abstinence) - the lifestyle of the female should be such that there is complete abstinence from intercourse from two weeks prior to the study until at least 72 hours after the end of the study , implants, injectables, combined oral contraceptives, hormonal IUDs, or double-barrier methods, i.e. any double combination of IUD, condom with spermicidal gel, diaphragm, sponge, and cervical cap)
6. Available to complete all study measurements

Exclusion Criteria:

1. History of lower respiratory tract infection four weeks prior to the informed consent visit
2. Past or present disease, which as judged by the investigator, may affect the outcome of this study. These diseases include, but are not limited to, cardiovascular disease, malignancy, hepatic disease, renal disease, hematological disease, neurological disease, endocrine disease or pulmonary disease (including but not confined to tuberculosis, bronchiectasis or cystic fibrosis)
3. History of drug or alcohol abuse
4. Suspected inability to understand the protocol requirements, instructions and study-related restrictions, the nature, scope, and possible consequences of the study
5. Inability to abstain from bronchodilators according to section 8.2 (Prohibited medication)
6. Risk of non-compliance with study procedures

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2010-03; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Characterization of particles in exhaled breath of subjects with COPD compared with healthy smokers. | within one day
  At visit 2, the exhaled particle analysis will be performed. These measurements will be repeated after 2 hours on the same day.
  Visit 3:
  After a baseline exhaled particle analysis, the subjects will inhale nebulized saline (2.5 ml of a 0.9 % NaCl-solution). Aerosol generation and transport will be recorded immediately after the end of inhalation as well as 2 hours and 4 hours.

CONTACTS AND LOCATIONS:
Overall Officials: Jens Hohlfeld, Prof. Dr., Principal Investigator — Fraunhofer Institute for Toxicology and Experimental Medicine
Locations (1):
- Fraunhofer Institute for Toxicolocy, Hanover, Lower Saxony, Germany

REFERENCES:
- See also: Related Info — http://www.atemwegsforschung.de